CLINICAL TRIAL: NCT01260324
Title: The Detection and Epidemiology of NAION in a Commercially Insured Population in the United States.
Brief Title: Epidemiology Study of Non-arteritic Anterior Ischemic Optic Neuropathy (NAION)
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A1481282
Record Dates: First submitted 2010-11-05; First posted 2010-12-15 (Estimated); Results first posted 2011-04-25 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Anterior Ischemic Optic Neuropathy; Ischemic Optic Neuropathy
Keywords: Phosphodiesterase type 5 inhibitors; non-arteritic anterior ischemic optic neuropathy; descriptive epidemiology study
MeSH Terms: conditions — Optic Neuropathy, Ischemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NAION cases: From the study population, patients with a claim associated with an ischemic optic neuropathy diagnosis code were identified as potential NAION cases (n = 3,732). From the potential NAION cases, definite and possible NAION cases were identified using medical record review and a claims algorithm (n=1,283). Data from definite and possible NAION cases contributed to the analysis.
  Interventions: Other: No intervention given in this observational study
- Controls: From the study population, patients without a claim associated with an ischemic optic neuropathy diagnosis code were randomly selected as controls (n = 20,000)
  Interventions: Other: No intervention given in this observational study

INTERVENTIONS:
Other: No intervention given in this observational study — No intervention given in this observational study
  Groups: NAION cases
Other: No intervention given in this observational study — No intervention given in this observational study
  Groups: Controls

SUMMARY:
The objectives of this study were to: (1) evaluate the natural history of non-arteritic anterior ischemic optic neuropathy (NAION); (2) estimate the population incidence of NAION; and (3) identify potential risk factors for NAION.

DETAILED DESCRIPTION:
The study population consisted of members of the Ingenix Normative Health Informatics (NHI) Database during 01/01/2003 through 12/31/2007, who were 18 years of age or older with at least 183 days of continuous enrollment in the database and without any doctor visits associated with a diagnosis of ischemic optic neuropathy during the 183 days prior to cohort entry.

From the study population, patients with a claim associated with an ischemic optic neuropathy diagnosis code were identified as potential NAION cases (n = 3,732). From the potential NAION cases, definite and possible NAION cases were identified using medical record review and a claims algorithm (n=1,283).

From the study population, patients without a claim associated with an ischemic optic neuropathy diagnosis code were randomly selected as controls (n = 20,000)

ELIGIBILITY:
Inclusion Criteria:

* Member of the Ingenix Normative Health Informatics (NHI) Database during 01/01/2003 through 12/31/2007
* 18 years of age or older
* Had at least 183 days of continuous enrollment in the database
* No doctor visits associated with a diagnosis of ischemic optic neuropathy during the 183 days prior to cohort entry

Exclusion Criteria:

* Less than 18 years of age
* Less than 183 days of continuous enrollment in the database
* At least one doctor visit associated with a diagnosis of ischemic optic neuropathy during the 183 days prior to cohort entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of members of the Ingenix Normative Health Informatics (NHI) Database during 01/01/2003 through 12/31/2007, who were 18 years of age or older with at least 183 days of continuous enrollment in the database and without any doctor visits associated with a diagnosis of ischemic optic neuropathy during the 183 days prior to cohort entry.
Sampling Method: Non-Probability Sample
Enrollment: 21283 (Actual)
Dates: Start 2008-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481282&StudyName=Epidemiology%20Study%20of%20Non-arteritic%20Anterior%20Ischemic%20Optic%20Neuropathy%20%28NAION%29

RESULTS

PARTICIPANT FLOW:
Groups:
- NAION Cases: Nonarteritic anterior ischemic optic neuropathy (NAION). From the study population, patients with a claim associated with an ischemic optic neuropathy diagnosis code were identified as potential NAION cases (n = 3,732). From the potential NAION cases, definite and possible NAION cases were identified using medical record review and a claims algorithm (n=1,283). Data from definite and possible NAION cases contributed to the analysis.
Period: Overall Study
Arm/Group | NAION Cases | Controls
Started | 1283 | 20000
Completed | 1283 | 20000
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NAION Cases | Controls | Total
Number analyzed (Participants) | 1283 | 20000 | 21283
Age, Customized [Number; unit: participants]
  18 to 34 years | 43 | 5954 | 5997
  35 to 44 years | 59 | 4937 | 4996
  45 to 54 years | 208 | 4655 | 4863
  55 to 64 years | 481 | 3041 | 3522
  65 to 74 years | 247 | 902 | 1149
  ≥75 years | 245 | 511 | 756
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 595 | 10669 | 11264
  Male | 688 | 9331 | 10019
Number of participants with NAION diagnosis per calendar year [Number; unit: participants] — Medical record-adjudicated definite and possible cases and claims algorithm-derived definite and possible cases.
  participants
    Year 2003 | 285 | 3953 | 4238
    Year 2004 | 236 | 3990 | 4226
    Year 2005 | 284 | 4137 | 4421
    Year 2006 | 231 | 4081 | 4312
    Year 2007 | 247 | 3839 | 4086
Number of participants with NAION diagnosis per region of United States [Number; unit: participants] — Medical record-adjudicated definite and possible cases and claims algorithm-derived definite and possible cases.
  participants
    Northeast | 100 | 2456 | 2556
    Midwest | 362 | 5345 | 5707
    South | 656 | 9158 | 9814
    West | 165 | 3041 | 3206

OUTCOME MEASURES:

1. Primary Outcome: Crude Incidence Rate of Non-arteritic Anterior Ischemic Optic Neuropathy (NAION) Per 1000 Person-years by Age
Description: Person-years estimated by dividing the number of Controls participants by the derived sampling fraction (20,000 divided by the total person-time at risk). Age categorized by years.
Time Frame: 01-January-2003 up to 31-December-2007
Population: Combined NAION cases and Controls populations; (n)=number of participants for NAION cases and Controls, respectively, per estimated person-years [(NAION cases n, Controls n) / person-years].
Measure: Number (95% Confidence Interval); unit: incidence rate per 1000 person-years
Groups:
- Combined NAION Cases and Controls: NAION cases: from the study population, patients with a claim associated with an ischemic optic neuropathy diagnosis code were identified as potential NAION cases (n = 3,732). From the potential NAION cases, definite and possible NAION cases were identified using medical record review and a claims algorithm (n=1,283). Data from definite and possible NAION cases contributed to the analysis.
  Controls: from the study population, patients without a claim associated with an ischemic optic neuropathy diagnosis code were randomly selected as controls (n = 20,000).
Arm/Group | Combined NAION Cases and Controls
Number analyzed (Participants) | 21283
incidence rate per 1000 person-years
  Age 18 to 34 (n=43, 5,954) / 8,042,997 | 0.01 [0.00 to 0.01]
  Age 35 to 44 (n=59, 4,937) / 6,669,176 | 0.01 [0.01 to 0.01]
  Age 45 to 54 (n=208, 4,655) / 6,288,235 | 0.03 [0.03 to 0.04]
  Age 55 to 64 (n=481, 3,041) / 4,107,953 | 0.12 [0.11 to 0.13]
  Age 65 to 74 (n=247, 902) / 1,218,472 | 0.20 [0.18 to 0.23]
  Age ≥75 (n=245, 511) / 690,287 | 0.35 [0.31 to 0.40]
Statistical Analysis 1: Comparison: Combined NAION Cases and Controls; Incidence rate Age 18 to 34; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.01, 95% CI 2-sided [0.01 to 0.01] — Standardized to the quintiles of the probability of having NAION predicted by all the other risk factors of NAION among the Controls
Statistical Analysis 2: Comparison: Combined NAION Cases and Controls; Incidence rate Age 35 to 44; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.01, 95% CI 2-sided [0.01 to 0.01] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Combined NAION Cases and Controls; Incidence rate Age 45 to 54; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.03, 95% CI 2-sided [0.03 to 0.04] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Combined NAION Cases and Controls; Incidence rate Age 55 to 64; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.08, 95% CI 2-sided [0.07 to 0.09] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Combined NAION Cases and Controls; Incidence rate Age 65 to 74; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.12, 95% CI 2-sided [0.11 to 0.14] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Combined NAION Cases and Controls; Incidence rate Age ≥75; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.18, 95% CI 2-sided [0.15 to 0.21] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Combined NAION Cases and Controls; Odds ratio Age 18 to 34; Test type: Superiority or Other; Odds Ratio (OR) = 0.09, 95% CI 2-sided [0.06 to 0.13] — Odds ratio derived from covariate-adjusted logisitic regression model and adjusted for all other covariates in the table
Statistical Analysis 8: Comparison: Combined NAION Cases and Controls; Odds ratio Age 35 to 44; Test type: Superiority or Other; Odds Ratio (OR) = 0.11, 95% CI 2-sided [0.08 to 0.16] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 9: Comparison: Combined NAION Cases and Controls; Odds ratio Age 45 to 54; Test type: Superiority or Other; Odds Ratio (OR) = 0.37, 95% CI 2-sided [0.30 to 0.45] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 10: Comparison: Combined NAION Cases and Controls; Odds ratio Age 65 to 74; Test type: Superiority or Other; Odds Ratio (OR) = 3.83, 95% CI 2-sided [2.68 to 5.47] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 11: Comparison: Combined NAION Cases and Controls; Odds ratio Age ≥75; Test type: Superiority or Other; Odds Ratio (OR) = 5.73, 95% CI 2-sided [4.00 to 8.22] — [estimate comment as in outcome 1, analysis 7]

2. Primary Outcome: Crude Incidence Rate of Non-arteritic Anterior Ischemic Optic Neuropathy (NAION) Per 1000 Person-years by Sex
Description: Person-years estimated by dividing the number of Controls participants by the derived sampling fraction (20,000 divided by the total person-time at risk). Sex categorized as Female or Male.
Time Frame: 01-January-2003 up to 31-December-2007
Population: Combined population includes NAION cases and Controls population; (n)=number of participants for NAION cases and Controls, respectively, and estimated person-years [(n=NAION cases, Controls) / person-years].
Measure: Number (95% Confidence Interval); unit: incidence rate per 1000 person-years
Arm/Group | Combined NAION Cases and Controls
Number analyzed (Participants) | 21283
incidence rate per 1000 person-years
  Female (n=595, 10,669) / 14,412,283 | 0.04 [0.04 to 0.04]
  Male (n=688, 9,331) / 12,604,837 | 0.05 [0.05 to 0.06]
Statistical Analysis 1: Comparison: Combined NAION Cases and Controls; Incidence rate Female; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.04, 95% CI 2-sided [0.04 to 0.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Combined NAION Cases and Controls; Incidence rate Male; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.05, 95% CI 2-sided [0.05 to 0.06] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Combined NAION Cases and Controls; Odds ratio Male; Test type: Superiority or Other; Odds Ratio (OR) = 1.83, 95% CI 2-sided [1.50 to 2.22] — [estimate comment as in outcome 1, analysis 7]

3. Primary Outcome: Crude Incidence Rate of Non-arteritic Anterior Ischemic Optic Neuropathy (NAION) Per 1000 Person-years by Calendar Year
Description: Person-years estimated by dividing the number of Controls participants by the derived sampling fraction (20,000 divided by the total person-time at risk). Calendar years include years 2003 to 2007.
Time Frame: 01-January-2003 up to 31-December-2007
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: incidence rate per 1000 person-years
Arm/Group | Combined NAION Cases and Controls
Number analyzed (Participants) | 21283
incidence rate per 1000 person-years
  Year 2003 (n=285, 3953) / 5,339,934 | 0.05 [0.05 to 0.06]
  Year 2004 (n=236, 3,990) / 5,389,915 | 0.04 [0.04 to 0.05]
  Year 2005 (n=284, 4,137) / 5,588,491 | 0.05 [0.05 to 0.06]
  Year 2006 (n=231, 4,081) / 5,512,843 | 0.04 [0.04 to 0.05]
  Year 2007 (n=247, 3,839) / 5,185,936 | 0.05 [0.04 to 0.05]
Statistical Analysis 1: Comparison: Combined NAION Cases and Controls; Incidence rate Year 2003; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.05, 95% CI 2-sided [0.04 to 0.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Combined NAION Cases and Controls; Incidence rate Year 2004; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.05, 95% CI 2-sided [0.04 to 0.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Combined NAION Cases and Controls; Incidence rate Year 2005; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.05, 95% CI 2-sided [0.04 to 0.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Combined NAION Cases and Controls; Incidence rate Year 2006; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.04, 95% CI 2-sided [0.04 to 0.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Combined NAION Cases and Controls; Incidence rate Year 2007; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.05, 95% CI 2-sided [0.04 to 0.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Combined NAION Cases and Controls; Odds ratio Year 2004; Test type: Superiority or Other; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.61 to 0.96] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 7: Comparison: Combined NAION Cases and Controls; Odds ratio Year 2005; Test type: Superiority or Other; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.58 to 0.91] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 8: Comparison: Combined NAION Cases and Controls; Odds ratio Year 2006; Test type: Superiority or Other; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.68 to 1.12] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 9: Comparison: Combined NAION Cases and Controls; Odds ratio Year 2007; Test type: Superiority or Other; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.72 to 1.19] — [estimate comment as in outcome 1, analysis 7]

4. Primary Outcome: Crude Incidence Rate of Non-arteritic Anterior Ischemic Optic Neuropathy (NAION) Per 1000 Person-years by Region
Description: Person-years estimated by dividing the number of Controls participants by the derived sampling fraction (20,000 divided by the total person-time at risk). Region of the United States categorized as Northeast, Midwest, South, and West.
Time Frame: 01-January-2003 up to 31-December-2007
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: incidence rate per 1000 person-years
Arm/Group | Combined NAION Cases and Controls
Number analyzed (Participants) | 21283
incidence rate per 1000 person-years
  Northeast (n=100, 2,456) / 3,317,702 | 0.03 [0.02 to 0.04]
  Midwest (n=362, 5,345) / 7,220,325 | 0.05 [0.05 to 0.06]
  South (n=656, 9,158) / 12,371,139 | 0.05 [0.05 to 0.06]
  West (n=165, 3,041) / 4,107,953 | 0.04 [0.03 to 0.05]
Statistical Analysis 1: Comparison: Combined NAION Cases and Controls; Incidence rate Northeast; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.05, 95% CI 2-sided [0.04 to 0.06] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Combined NAION Cases and Controls; Incidence rate Midwest; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.05, 95% CI 2-sided [0.04 to 0.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Combined NAION Cases and Controls; Incidence rate South; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.05, 95% CI 2-sided [0.05 to 0.06] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Combined NAION Cases and Controls; Incidence rate West; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.04, 95% CI 2-sided [0.04 to 0.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Combined NAION Cases and Controls; Odds ratio Northeast; Test type: Superiority or Other; Odds Ratio (OR) = 0.41, 95% CI 2-sided [0.31 to 0.56] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 6: Comparison: Combined NAION Cases and Controls; Odds ratio Midwest; Test type: Superiority or Other; Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.56 to 0.84] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 7: Comparison: Combined NAION Cases and Controls; Odds ratio West; Test type: Superiority or Other; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.57 to 0.93] — [estimate comment as in outcome 1, analysis 7]

5. Primary Outcome: Crude Incidence Rate of Non-arteritic Anterior Ischemic Optic Neuropathy (NAION) Per 1000 Person-years by Baseline Risk Factors
Description: Person-years estimated by dividing number of Controls (20,000) by derived sampling fraction (total person-time at risk). Risk factors include diabetes, smoking, obesity, erectile dysfunction, hyperlipidemia, myocardial infarction, other coronary artery disease, congestive heart failure, hypertension, use of beta or calcium channel blockers, angiotensin-converting enzyme inhibitors, nitrates, anti-platelet agents, diuretics, and recent phosphodiesterase type 5 (PDE-5) inhibitors use. Recent use=any dispensing in the 60 days preceding date of diagnosis for NAION cases or index date for Controls.
Time Frame: 01-January-2003 up to 31-December-2007
Population: Combined population; (n)=number of participants for NAION cases and Controls, respectively, and estimated person-years [(n=NAION cases, Controls) / person-years]. Only the covariates selected by the step wise regression procedure were summarized.
Measure: Number (95% Confidence Interval); unit: incidence rate per 1000 person-years
Arm/Group | Combined NAION Cases and Controls
Number analyzed (Participants) | 21283
incidence rate per 1000 person-years
  Diabetes (n=349, 1,131) / 1,527,818 | 0.23 [0.21 to 0.25]
  Smoking (n=48, 232) / 313,399 | 0.15 [0.11 to 0.20]
  Obesity (n=25, 273) / 368,784 | 0.07 [0.04 to 0.10]
  Nitrates (n=71, 171) / 230,996 | 0.31 [0.24 to 0.39]
  Anti-platelet agents (n=127, 182) / 245,856 | 0.52 [0.43 to 0.61]
  Diuretics (n=134, 296) / 399,853 | 0.34 [0.28 to 0.40]
  Recent PDE-5 inhibitors use (n=17, 202) / 272,873 | 0.06 [0.04 to 0.10]
Statistical Analysis 1: Comparison: Combined NAION Cases and Controls; Incidence rate Diabetes; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.09, 95% CI 2-sided [0.08 to 0.10] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Combined NAION Cases and Controls; Incidence rate Smoking; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.11, 95% CI 2-sided [0.08 to 0.14] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Combined NAION Cases and Controls; Incidence rate Obesity; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.04, 95% CI 2-sided [0.03 to 0.06] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Combined NAION Cases and Controls; Incidence rate Nitrates; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.07, 95% CI 2-sided [0.06 to 0.09] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Combined NAION Cases and Controls; Incidence rate Anti-platelet agents; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.15, 95% CI 2-sided [0.12 to 0.18] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Combined NAION Cases and Controls; Incidence rate Diuretics; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.13, 95% CI 2-sided [0.09 to 0.17] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Combined NAION Cases and Controls; Incidence rate Recent PDE-5 inhibitors use; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.03, 95% CI 2-sided [0.01 to 0.04] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Combined NAION Cases and Controls; Odds ratio Diabetes; Test type: Superiority or Other; Odds Ratio (OR) = 1.82, 95% CI 2-sided [1.47 to 2.25] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 9: Comparison: Combined NAION Cases and Controls; Odds ratio Smoking; Test type: Superiority or Other; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.63 to 2.85] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 10: Comparison: Combined NAION Cases and Controls; Odds ratio Obesity; Test type: Superiority or Other; Odds Ratio (OR) = 0.43, 95% CI 2-sided [0.23 to 0.81] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 11: Comparison: Combined NAION Cases and Controls; Odds ratio Nitrates; Test type: Superiority or Other; Odds Ratio (OR) = 0.63, 95% CI 2-sided [0.42 to 0.94] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 12: Comparison: Combined NAION Cases and Controls; Odds ratio Anti-platelet agents; Test type: Superiority or Other; Odds Ratio (OR) = 2.12, 95% CI 2-sided [1.53 to 2.94] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 13: Comparison: Combined NAION Cases and Controls; Odds ratio Diuretics; Test type: Superiority or Other; Odds Ratio (OR) = 2.24, 95% CI 2-sided [1.46 to 3.43] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 14: Comparison: Combined NAION Cases and Controls; Odds ratio Recent PDE-5 inhibitors use; Test type: Superiority or Other; Odds Ratio (OR) = 0.57, 95% CI 2-sided [0.31 to 1.04] — [estimate comment as in outcome 1, analysis 7]

6. Primary Outcome: Crude Incidence Rate of Non-arteritic Anterior Ischemic Optic Neuropathy (NAION) Per 1000 Person-years by Comorbid Diagnoses
Description: Person-years estimated by dividing the number of Controls participants by the derived sampling fraction (20,000 divided by the total person-time at risk). Comorbid diagnoses categorized according to the International Classification of Diseases ninth-edition (ICD-9) diagnoses. Categories include Occlusion and stenosis of precerebral arteries (Occlusion / Stenosis), Other disorders of bone and cartilage (Bone and Cartilage), Symptoms involving head and neck (Head and Neck), and Other ill defined and unknown causes of morbidity and mortality (Ill defined / Unknown causes).
Time Frame: 01-January-2003 up to 31-December-2007
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: incidence rate per 1000 person-years
Arm/Group | Combined NAION Cases and Controls
Number analyzed (Participants) | 21283
incidence rate per 1000 person-years
  Other retinal disorders (n=337, 240) / 324,205 | 1.04 [0.93 to 1.16]
  Glaucoma (n=161, 353) / 476,852 | 0.34 [0.29 to 0.39]
  Cataract (n=245, 405) / 547,097 | 0.45 [0.39 to 0.51]
  Visual disturbances (n=291, 130) / 175,611 | 1.66 [1.47 to 1.86]
  Blindness and low vision (n=103, 11) / 14,859 | 6.93 [5.66 to 8.41]
  Other disorders of eye (n=143, 201) / 271,522 | 0.53 [0.44 to 0.62]
  Occlusion / Stenosis (n=98, 75) / 101,314 | 0.97 [0.79 to 1.18]
  Acute sinusitis (n=92, 1,123) / 1,517,011 | 0.06 [0.05 to 0.07]
  Other dermatoses (n=114, 536) / 724,059 | 0.16 [0.13 to 0.19]
  Bone and cartilage (n=114, 504) / 680,831 | 0.17 [0.14 to 0.20]
  Head and neck (n=181, 771) / 1,041,510 | 0.17 [0.15 to 0.20]
  Ill defined / Unknown causes (n=71, 183) / 247,207 | 0.29 [0.22 to 0.36]
Statistical Analysis 1: Comparison: Combined NAION Cases and Controls; Incidence rate Other retinal disorders; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.33, 95% CI 2-sided [0.28 to 0.39] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Combined NAION Cases and Controls; Incidence rate Glaucoma; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.13, 95% CI 2-sided [0.11 to 0.16] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Combined NAION Cases and Controls; Incidence rate Cataract; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.20, 95% CI 2-sided [0.08 to 0.41] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Combined NAION Cases and Controls; Incidence rate Visual disturbances; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.99, 95% CI 2-sided [0.83 to 1.17] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Combined NAION Cases and Controls; Incidence rate Blindness and low vision; Test type: Superiority or Other; Incidence rate per 1000 person-years = 2.00, 95% CI 2-sided [1.60 to 2.46] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Combined NAION Cases and Controls; Incidence rate Other disorders of eye; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.19, 95% CI 2-sided [0.16 to 0.23] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Combined NAION Cases and Controls; Incidence rate Occlusion and stenosis of precerebral arteries; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.22, 95% CI 2-sided [0.18 to 0.27] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Combined NAION Cases and Controls; Incidence rate Acute sinusitis; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.07, 95% CI 2-sided [0.05 to 0.08] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Combined NAION Cases and Controls; Incidence rate Other dermatoses; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.06, 95% CI 2-sided [0.05 to 0.08] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Combined NAION Cases and Controls; Incidence rate Other disorders of bone and cartilage; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.08, 95% CI 2-sided [0.06 to 0.10] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Combined NAION Cases and Controls; Incidence rate Symptoms involving head and neck; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.12, 95% CI 2-sided [0.10 to 0.14] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Combined NAION Cases and Controls; Incidence rate Other ill defined and unknown causes of morbidity and mortality; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.14, 95% CI 2-sided [0.10 to 0.18] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Combined NAION Cases and Controls; Odds ratio Other retinal disorders; Test type: Superiority or Other; Odds Ratio (OR) = 6.65, 95% CI 2-sided [4.72 to 9.38] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 14: Comparison: Combined NAION Cases and Controls; Odds ratio Glaucoma; Test type: Superiority or Other; Odds Ratio (OR) = 2.60, 95% CI 2-sided [1.77 to 3.81] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 15: Comparison: Combined NAION Cases and Controls; Odds ratio Cataract; Test type: Superiority or Other; Odds Ratio (OR) = 1.31, 95% CI 2-sided [1.02 to 1.68] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 16: Comparison: Combined NAION Cases and Controls; Odds ratio Visual disturbances; Test type: Superiority or Other; Odds Ratio (OR) = 14.20, 95% CI 2-sided [10.40 to 19.30] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 17: Comparison: Combined NAION Cases and Controls; Odds ratio Blindness and low vision; Test type: Superiority or Other; Odds Ratio (OR) = 15.10, 95% CI 2-sided [6.60 to 34.50] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 18: Comparison: Combined NAION Cases and Controls; Odds ratio Other disorders of eye; Test type: Superiority or Other; Odds Ratio (OR) = 2.02, 95% CI 2-sided [1.44 to 2.82] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 19: Comparison: Combined NAION Cases and Controls; Odds ratio Occlusion and stenosis of precerebral arteries; Test type: Superiority or Other; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.64 to 2.31] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 20: Comparison: Combined NAION Cases and Controls; Odds ratio Acute sinusitis; Test type: Superiority or Other; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.96 to 1.74] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 21: Comparison: Combined NAION Cases and Controls; Odds ratio Other dermatoses; Test type: Superiority or Other; Odds Ratio (OR) = 1.34, 95% CI 2-sided [1.02 to 1.77] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 22: Comparison: Combined NAION Cases and Controls; Odds ratio Other disorders of bone and cartilage; Test type: Superiority or Other; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.98 to 1.77] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 23: Comparison: Combined NAION Cases and Controls; Odds ratio Symptoms involving head and neck; Test type: Superiority or Other; Odds Ratio (OR) = 1.37, 95% CI 2-sided [1.02 to 1.84] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 24: Comparison: Combined NAION Cases and Controls; Odds ratio Ill defined and unknown causes of morbidity and mortality; Test type: Superiority or Other; Odds Ratio (OR) = 1.64, 95% CI 2-sided [1.08 to 2.49] — [estimate comment as in outcome 1, analysis 7]

7. Primary Outcome: Crude Incidence Rate of Non-arteritic Anterior Ischemic Optic Neuropathy (NAION) Per 1000 Person-years by PDE-5 Inhibitor Use
Description: Person-years estimated by dividing the number of Controls by the derived sampling fraction (20,000 divided by total person-time at risk). PDE-5 inhibitor use categorized by frequency of use in the number of days specific preceding diagnosis for NAION Cases or preceding the index date for Controls: Recent use=any dispensing in the preceding 60 days; Any use=any PDE-5 inhibitors use; Chronic use=at least a total of 26 days supply or 5 dispensings in the preceding 183 days; Non-chronic use=any dispensing in the preceding 183 days that does not meet the criteria for chronic use; Never use=none.
Time Frame: 01-January-2003 up to 31-December-2007
Population: Combined NAION cases and Controls populations. N=number of participants according to frequency of PDE-5 inhibitor use for males 40 years or older; (n)=number of participants for NAION cases and Controls, respectively, per variable of frequency of use and estimated person-years [(n=NAION cases, Controls) / person-years].
Measure: Number (95% Confidence Interval); unit: incidence rate per 1000 person-years
Arm/Group | Combined NAION Cases and Controls
Number analyzed (Participants) | 6219
incidence rate per 1000 person-years
  Recent use (n=17, 187) / 254,239 | 0.05 [0.03 to 0.09]
  Any use (n=32, 322) / 437,780 | 0.06 [0.04 to 0.09]
  Chronic use (n=16, 162) / 220,249 | 0.06 [0.03 to 0.10]
  Non-chronic use (n=16, 160) / 217,530 | 0.07 [0.04 to 0.11]
  Never use (n=631, 5,234) / 7,115,962 | 0.09 [0.08 to 0.10]
Statistical Analysis 1: Comparison: Combined NAION Cases and Controls; Incidence rate Recent use; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.05, 95% CI 2-sided [0.03 to 0.07] — Standardized to the quintiles of the probability predicted by all the other risk factors of NAION among the Controls
Statistical Analysis 2: Comparison: Combined NAION Cases and Controls; Incidence rate Any use (includes chronic and non-chronic use); Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.06, 95% CI 2-sided [0.04 to 0.08] — Standardized to the quintiles of the probability predicted by all the other risk factors of NAION among the Controls
Statistical Analysis 3: Comparison: Combined NAION Cases and Controls; Incidence rate Chronic use; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.05, 95% CI 2-sided [0.03 to 0.08] — Standardized to the quintiles of the probability predicted by all the other risk factors of NAION among the Controls
Statistical Analysis 4: Comparison: Combined NAION Cases and Controls; Incidence rate Non-chronic use; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.06, 95% CI 2-sided [0.03 to 0.11] — Standardized to the quintiles of the probability predicted by all the other risk factors of NAION among the Controls
Statistical Analysis 5: Comparison: Combined NAION Cases and Controls; Incidence rate Never use; Test type: Superiority or Other; Incidence rate per 1000 person-years = 0.09, 95% CI 2-sided [0.08 to 0.10] — Standardized to the quintiles of the probability predicted by all the other risk factors of NAION among the Controls

8. Primary Outcome: Number of Participants With NAION by Time Course of Visual Change Onset: Intermittent, Abrupt (Acute), or Chronic (Adjudicated by Medical Record Review)
Time Frame: 01-January-2003 up to 31-December-2007
Population: Participants from the NAION cases population adjudicated by medical record review.
Measure: Number; unit: participants
Groups:
- NAION Cases: NAION cases: from the study population, patients with a claim associated with an ischemic optic neuropathy diagnosis code were identified as potential NAION cases (n = 3,732). From the potential NAION cases, definite and possible NAION cases were identified using medical record review. Data from definite and possible NAION cases identified from medical record review only contributed to the analysis.
Arm/Group | NAION Cases
Number analyzed (Participants) | 74
participants
  Acute | 35
  Intermittent | 3
  Chronic | 1
  Unknown | 35

9. Primary Outcome: Incidence Rate Ratio Between NAION Risk Factors and Resolution of Visual Symptoms of Non-arteritic Anterior Ischemic Optic Neuropathy (NAION)
Description: Categorized by risk factors of age (years) and sex (male or female). Incidence rate ratio and the 95% confidence interval adjusted for all the other covariates in the table.
Time Frame: 01-January-2003 up to 31-December-2007
Population: Participant population with definite and possible NAION cases identified by medical record review. N=number of participants with resolution of visual symptoms (each set of variables); (n)=number of participants for variable (age or sex) for NAION cases and estimated person-years [(n=NAION cases) / person-years].
Measure: Number (95% Confidence Interval); unit: incidence rate ratio
Arm/Group | NAION Cases
Number analyzed (Participants) | 57
incidence rate ratio
  Age 18 to 64 years (n=18) / 25.53 | 1.00 [NA to NA] — Result value is the reference category for calculation of the rate ratio; CI not applicable.
  Age ≥65 years (n=9) / 29.94 | 0.56 [0.25 to 1.25]
  Female (n=14) / 31.69 | 1.00 [NA to NA] — Result value is the reference category for calculation of the rate ratio; CI not applicable.
  Male (n=13) / 23.77 | 1.22 [0.57 to 2.62]

10. Primary Outcome: Incidence Rate Ratio Between NAION Risk Factors and Recurrence of Visual Symptoms of Non-arteritic Anterior Ischemic Optic Neuropathy (NAION)
Description: as for outcome 9
Time Frame: 01-January-2003 up to 31-December-2007
Population: Participant population with definite and possible NAION cases identified by medical record review. N=number of participants with recurrence of visual symptoms; (n)=number of participants for variable (age or sex) for NAION cases and estimated person-years [(n=NAION cases) / person-years].
Measure: Number (95% Confidence Interval); unit: incidence rate ratio
Arm/Group | NAION Cases
Number analyzed (Participants) | 74
incidence rate ratio
  Age 18 to 64 years (n=2) / 66.63 | 1.00 [NA to NA] — Result value is the reference category for calculation of the rate ratio; CI not applicable.
  Age ≥65 years (n=1) / 57.39 | 0.62 [0.06 to 6.96]
  Female (n=1) / 66.05 | 1.00 [NA to NA] — Result value is the reference category for calculation of the rate ratio; CI not applicable.
  Male (n=2) / 57.97 | 2.03 [0.18 to 22.70]

ADVERSE EVENTS:
Time Frame: 1-January-2003 up to 31-December-2007
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | NAION Cases | Controls
Serious Adverse Events (participants affected / at risk) | 0/1283 | 0/20000
Other Adverse Events (participants affected / at risk) | 0/1283 | 0/20000

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.